CLINICAL TRIAL: NCT02253589
Title: Evaluation of Motivational Interviewing (MI) to Reduce Khat Use Among Somali Refugees in Kenya
Brief Title: Motivational Interviewing (MI) to Reduce Khat Use
Acronym: MIkhat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Researcher, University of Konstanz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01DG13020
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Khat Use Disorder
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list (No Intervention): Participants will assessment only during study, same intervention after posttest
- Intervention (Experimental): Participants assigned to this arm will receive the modified ASSIST-linked Brief Intervention
  Interventions: Behavioral: modified ASSIST-linked Brief Intervention

INTERVENTIONS:
Behavioral: modified ASSIST-linked Brief Intervention — Trained counsellors support participant's motivation to reduce or stop khat use in a 20 minute counselling session.
  Other Names: Motivational Interviewing
  Arms: Intervention

SUMMARY:
Healthy khat user with the intention to reduce or stop khat use will be randomly assigned to a one-session brief intervention or waiting list. Reductions in khat use will be measured from pre- to post-assessment which will be one month apart. After one month, the waiting list will receive the same intervention.

DETAILED DESCRIPTION:
The leaves of the khat tree are traditionally chewed in some African and Arab countries. They contain the mild central stimulant cathinone. In recent years, the production, trade and use has dramatically increased and excessive patterns of use as well as a specific dependence syndrome have been described. So far, no experiences exist in psychological treatment of khat addiction.

In this study, we use a brief motivational intervention based on the WHO's ASSIST-linked Brief Intervention and Motivational Interviewing to support users who have the intention to reduce or stop their khat use. Khat users will be recruited in the community. Trained local staff will assess participant's khat and other substance use at study entry and one month later. Users will be assigned randomly to intervention or waiting list control groups. The intervention group will receive a single 20-minute brief intervention. The waiting list will receive the same intervention after the second assessment. After two months, a final assessment will be made in both groups.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals

Exclusion Criteria:

Severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time-Line-Follow-Back: Self-reported days with khat use and amount of khat use | one month
  Participants report in a calender for each day of the past month whether they used khat and how much of it.

SECONDARY OUTCOMES:
Time-Line-Follow-Back: other substance use | One month
  Participants report for each day of the past month whether they used other substances of abuse, i.e. alcohol, illegal drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Tawakal Clinic, Nairobi, Kenya

REFERENCES:
- [Derived] Widmann M, Apondi B, Musau A, Warsame AH, Isse M, Mutiso V, Veltrup C, Schalinski I, Ndetei D, Odenwald M. Reducing Khat use among Somalis living in Kenya: a controlled pilot study on the modified ASSIST-linked brief intervention delivered in the community. BMC Public Health. 2022 Dec 5;22(1):2271. doi: 10.1186/s12889-022-14681-w. PMID 36471268